CLINICAL TRIAL: NCT00006237
Title: Phase III Trial of High Dose Interferon Alfa 2-b Versus Cisplatin, Vinblastine, DTIC Plus IL-2 and Interferon in Patients With High Risk Melanoma
Brief Title: S0008: Chemotherapy Plus Biological Therapy in Treating Patients With Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); Cancer and Leukemia Group B (Network); Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S0008; U10CA032102 (NIH); S0008 (Other: SWOG); CALGB-500002 (Other: CALGB); ECOG-S0008 (Other: ECOG); COG-S0008 (Other: COG); NCT00546416 (obsolete NCT alias)
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Results first posted 2012-09-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Interleukin-2; aldesleukin; Filgrastim; Interferon-alpha; Cisplatin; Dacarbazine; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Active Comparator): Patients receive interferon alfa IV on days 1-5 of weeks 1-4 followed by interferon alfa subcutaneously (SC) on days 1, 3, and 5 of weeks 5-52 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: interferon alfa
- Arm II (Experimental): Patients receive cisplatin IV over 30 minutes followed by vinblastine IV on days 1-4. Patients also receive dacarbazine IV over 1 hour on day 1, interleukin-2 IV over 96 hours on days 1-4, and interferon alfa SC on days 1-5, 8, 10, and 12. In addition, patients receive filgrastim (G-CSF) SC on days 6-15. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: interleukin-2; Biological: filgrastim; Biological: interferon alfa; Drug: cisplatin; Drug: dacarbazine; Drug: vinblastine

INTERVENTIONS:
Biological: interleukin-2 — Given IV
  Other Names: aldesleukin
  Arms: Arm II
Biological: filgrastim — Given subcutaneously
  Arms: Arm II
Biological: interferon alfa — Given IV and subcutaneously
Drug: cisplatin — Given IV
  Arms: Arm II
Drug: dacarbazine — Given IV
  Arms: Arm II
Drug: vinblastine — Given IV
  Arms: Arm II

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of cancer cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Interleukin-2 may stimulate a person's white blood cells to kill melanoma cells. It is not yet known whether interferon alfa is more effective with or without combination chemotherapy and interleukin-2 for melanoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of interferon alfa with or without combination chemotherapy consisting of cisplatin, vinblastine, and dacarbazine, plus interleukin-2, in treating patients who have melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival and disease-free survival of patients with high-risk melanoma treated with interferon alfa vs cisplatin, vinblastine, and dacarbazine plus interferon alfa and interleukin-2.
* Compare the toxic effects of these treatment regimens in these patients.
* Determine the relationship between minimal residual disease (MRD) status at 12 weeks and 52 weeks and overall survival of patients treated with these regimens.
* Compare the effects of these treatment regimens on the MRD status of these patients.
* Determine the relationship between clinical characteristics (number of involved lymph nodes, ulcerated primary, and extracapsular extension) and MRD in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to nodal status (N1 or N2 vs N3), degree of lymph node involvement (micrometastases only vs any macrometastases, including satellite/in-transit metastases), and ulceration of the primary tumor (yes vs no vs unknown primary). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive interferon alfa IV on days 1-5 of weeks 1-4 followed by interferon alfa subcutaneously (SC) on days 1, 3, and 5 of weeks 5-52 in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive cisplatin IV over 30 minutes followed by vinblastine IV on days 1-4. Patients also receive dacarbazine IV over 1 hour on day 1, interleukin-2 IV over 96 hours on days 1-4, and interferon alfa SC on days 1-5, 8, 10, and 12. In addition, patients receive filgrastim (G-CSF) SC on days 6-15. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually for 5 years.

PROJECTED ACCRUAL: A total of 410 patients (205 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven melanoma of cutaneous origin or from unknown primary at initial presentation of primary or first clinically detected nodal or satellite/in-transit recurrence

  * No distant metastases
  * No melanoma of ocular, mucosal, or other non-cutaneous origin
* One of the following criteria must apply for patients with newly diagnosed melanoma OR a previously diagnosed primary with current subsequent, clinical, regional nodal disease and/or satellite/in-transit disease:

  * Ulcerated primary melanoma with 1 or more involved lymph nodes (micro/occult or macro/clinically overt)
  * Non-ulcerated or unknown primary melanoma with one macro/clinically overt lymph node metastasis, including a single matted nodal mass

    * No non-ulcerated or unknown primary tumor and a single micrometastatic lymph node
  * Non-ulcerated melanoma with two or more lymph node metastases (micro/occult or macro/clinically overt) and/or matted nodes
  * Any satellite/in transit metastasis with or without lymph node involvement
* Patients with recurrent disease must have recurrent disease in the regional nodal basin of a prior complete lymphadenectomy
* Multiple regional nodal basin involvement allowed if they are appropriate anatomic drainage basins for primary site
* Patients must be disease free at time of enrollment based on the following surgical criteria:

  * Patients at initial presentation of melanoma must undergo adequate wide excision of primary lesion
  * Patients with previously diagnosed melanoma must have all disease resected with pathologically negative margins and no disease at primary site or second resection of primary
  * Full lymphadenectomy required of all patients including those with positive sentinel nodes or positive satellite/in-transit metastasis
* No more than 56 days since prior lymphadenectomy OR surgery to remove recurrent disease after prior complete lymphadenectomy
* Must be willing to participate in minimal residual disease studies if registered on the study on 3/1/2003 or later

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT or SGPT no greater than 2 times ULN
* LDH and alkaline phosphatase no greater than 2 times ULN (above normal value requires a contrast-enhanced CT scan or MRI of liver)
* No known recent hepatitis positivity by PCR

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 75 mL/min

Cardiovascular:

* No congestive heart failure
* No coronary artery disease
* No serious cardiac arrhythmia
* No prior myocardial infarction
* Normal cardiac stress test required if any of the following are present:

  * Over age 50
  * Abnormal EKG
  * History of cardiac disease

Pulmonary:

* No symptomatic pulmonary disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No autoimmune disorders or conditions of immunosuppression
* No other prior malignancy within the past 5 years except the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * Carcinoma in situ of the cervix
  * Adequately treated stage I or II cancer in remission
* HIV negative
* No known AIDS or HIV-1 associated complex

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy, including interferon, interleukin, levamisole, or other biologic response modifiers
* No other concurrent biologic therapy

Chemotherapy:

* No prior chemotherapy (including infusion or perfusion therapy)
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent systemic corticosteroids or topical steroid creams
* Concurrent steroid antihistamines allowed if no alternative
* No concurrent hormonal therapy

Radiotherapy:

* No prior radiotherapy

  * Prior postlumpectomy radiotherapy for breast cancer allowed
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* No concurrent surgery

Other:

* No concurrent anti-hypertensive medications (arm II only)
* No concurrent immunosuppressive agents
* No other concurrent anticancer therapy
* Antihistamines allowed if no alternative medication suitable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2000-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence E. Flaherty, MD, Study Chair — Barbara Ann Karmanos Cancer Institute; John A. Thompson, MD, Principal Investigator — Seattle Cancer Care Alliance; John T. Vetto, MD, FACS, Principal Investigator — OHSU Knight Cancer Institute; Michael B. Atkins, MD, Study Chair — Beth Israel Deaconess Medical Center; John M. Kirkwood, MD, Principal Investigator — University of Pittsburgh; Frank Haluska, MD, PhD, Study Chair — Massachusetts General Hospital; Alberto S. Pappo, MD, Principal Investigator — Texas Children's Cancer Center
Locations (297):
- United States (296):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Banner Thunderbird Medical Center, Glendale, Arizona
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Eden Medical Center, Castro Valley, California
  - Saint Rose Hospital, Hayward, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Valley Care Medical Center, Pleasanton, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - Scripps Cancer Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - CCOP - Santa Rosa Memorial Hospital, Sana Rosa, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Winship Cancer Institute of Emory University, Altanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago Westside Hospital, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Sherman Hospital, Elgin, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Hematology/Oncology of the North Shore at Gross Point Medical Center, Skokie, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Union Hospital Cancer Program at Union Hospital, Elkton MD, Maryland
  - Tufts-NEMC Cancer Center, Boston, Massachusetts
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Great Lakes Cancer Institute at McLaren Regional Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Upper Michigan Cancer Center at Marquette General Hospital, Marquette, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Booker Cancer Center at Riverview Medical Center, Red Bank, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Lovelace Medical Center - Gibson, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Adirondack Cancer Care - Glens Falls, Glens Falls, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Central Pennsylvania Hematology and Medical Oncology Associates, PC, Lemoyne, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee Cancer Institute - Memphis, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Martha Jefferson Hospital Cancer Care Center, Charlottesville, Virginia
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Fox Valley Hematology and Oncology - East Grant Street, Appleton, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia

REFERENCES:
- [Derived] Flaherty LE, Othus M, Atkins MB, Tuthill RJ, Thompson JA, Vetto JT, Haluska FG, Pappo AS, Sosman JA, Redman BG, Moon J, Ribas A, Kirkwood JM, Sondak VK. Southwest Oncology Group S0008: a phase III trial of high-dose interferon Alfa-2b versus cisplatin, vinblastine, and dacarbazine, plus interleukin-2 and interferon in patients with high-risk melanoma--an intergroup study of cancer and leukemia Group B, Children's Oncology Group, Eastern Cooperative Oncology Group, and Southwest Oncology Group. J Clin Oncol. 2014 Nov 20;32(33):3771-8. doi: 10.1200/JCO.2013.53.1590. Epub 2014 Oct 20. PMID 25332243

RESULTS

PARTICIPANT FLOW:
Groups:
- Interferon: interferon alfa IV
- Biochemotherapy: cisplatin, dacarbazine, interleukin-2, interferon alfa SC, filgrastim
Period: Overall Study
Arm/Group | Interferon | Biochemotherapy
Started | 212 | 220
Eligible | 203 | 200
Eligible and Treated | 203 | 199
Completed | 87 | 159
Not Completed | 125 | 61
Not completed — Adverse Event | 39 | 29
Not completed — Death | 1 | 0
Not completed — Refusal unrelated to adverse effects | 8 | 4
Not completed — Progression/relapse | 54 | 2
Not completed — Not eligible | 9 | 20
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Not protocol specified | 14 | 5

BASELINE CHARACTERISTICS:
Groups:
- Interferon: interferon alfa
- Total: Total of all reporting groups
Arm/Group | Interferon | Biochemotherapy | Total
Number analyzed (Participants) | 203 | 199 | 402
Age, Continuous [Median (Full Range); unit: years] | 47 [12 to 73] | 46 [10 to 74] | 47 [10 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 58 | 120
  Male | 141 | 141 | 282
Region of Enrollment [Number; unit: participants]
  United States | 203 | 199 | 402

OUTCOME MEASURES:

1. Primary Outcome: 5-year Overall Survival
Description: Overall survival was measured from the date of registration to study until death from any cause with observations censored at the date of last contact for patients last known to be alive.
Time Frame: Every three months for a year, every six months for years 2-5, annual for years 5-10
Measure: Number; unit: Percent of population
Groups:
- Interferon: interferon alfa IV on days 1-5 of weeks 1-4 followed by interferon alfa subcutaneously (SC) on days 1, 3, and 5 of weeks 5-52 in the absence of disease progression or unacceptable toxicity.
Arm/Group | Interferon | Biochemotherapy
Number analyzed (Participants) | 203 | 199
Percent of population | 56 | 56
Statistical Analysis 1: Comparison: Interferon vs Biochemotherapy; Test type: Superiority or Other; p = 0.49, Log Rank

2. Primary Outcome: 5-year Relapse-Free Survival
Description: Measured from date of registration to date of first observation of progressive disease or death due to any cause.
Time Frame: Every three months for the first year, every 6 months for years 2-5, annually for years 6-10
Measure: Number; unit: Percentage of population
Arm/Group | Interferon | Biochemotherapy
Number analyzed (Participants) | 203 | 199
Percentage of population | 47 | 38
Statistical Analysis 1: Comparison: Interferon vs Biochemotherapy; Test type: Superiority or Other; p = 0.02, Log Rank

3. Secondary Outcome: Toxicity
Description: Number of patients with Grade 3-5 adverse events that are related to study drug by given type of adverse event
Time Frame: While on treatment, patients on the HDIFN arm were assessed weekly for the 1st month, then every 2 weeks for the 2nd month, then every 3 months therafter; patients on the biochemo arm were assessed daily for the 1st 5 days, then weekly thereafter.
Population: Eligible patients who started therapy
Measure: Number; unit: Participants
Groups:
- Interferon: Interferon
- Biochemotherapy: Biochemotherapy
Arm/Group | Interferon | Biochemotherapy
Number analyzed (Participants) | 193 | 185
Participants
  Abdominal pain/cramping | 1 | 1
  Acidosis | 0 | 1
  Acute vascular leak syndrome | 0 | 1
  Alkaline phosphatase increase | 0 | 3
  Allergic reaction | 1 | 0
  Anal incontinence | 0 | 1
  Anemia | 0 | 8
  Anorexia | 1 | 9
  Anxiety/agitation | 4 | 5
  Apnea | 1 | 0
  Arrhythmia, NOS | 2 | 0
  Arthralgia | 4 | 3
  Bilirubin increase | 0 | 1
  Bone pain | 0 | 4
  CPK increase | 0 | 1
  Cardiovascular-other | 1 | 0
  Catheter related infection | 0 | 2
  Cerebrovascular ischemia | 1 | 0
  Colitis | 0 | 2
  Confusion | 2 | 3
  Constipation/bowel obstruction | 0 | 4
  Cranial neuropathy | 1 | 0
  Creatinine increase | 0 | 4
  Dehydration | 1 | 7
  Delusions | 0 | 1
  Depression | 14 | 4
  Diarrhea without colostomy | 2 | 6
  Dizziness/light headedness | 2 | 1
  Dizziness/vertigo, NOS | 0 | 1
  Double vision | 0 | 1
  Dyspnea | 1 | 2
  Eryth/rash/eruption/desq, NOS | 1 | 3
  Esophagitis/dysphagia | 0 | 2
  Eye-other | 1 | 0
  Fatigue/malaise/lethargy | 38 | 22
  Febrile neutropenia | 1 | 9
  Fever without neutropenia | 1 | 5
  Fever, NOS | 0 | 1
  Hallucinations | 1 | 1
  Headache | 9 | 5
  Hemorrhage w/ 3-4 thrombocyt | 0 | 1
  Hyperglycemia | 2 | 3
  Hyperkalemia | 0 | 1
  Hypermagnesemia | 1 | 1
  Hypertension | 0 | 1
  Hypertriglyceridemia | 1 | 0
  Hypocalcemia | 0 | 18
  Hypokalemia | 1 | 7
  Hypomagnesemia | 0 | 5
  Hyponatremia | 0 | 6
  Hypophosphatemia | 0 | 4
  Hypotension | 0 | 16
  Hypoxia | 0 | 1
  Infection w/o 3-4 neutropenia | 0 | 3
  Infection with 3-4 neutropenia | 0 | 9
  Infection, unk ANC | 1 | 2
  Insomnia | 1 | 1
  Leukopenia | 12 | 38
  Lipase increase | 1 | 2
  Local injection site reaction | 1 | 0
  Lymphopenia | 0 | 2
  Mood/consciousness change, NOS | 0 | 1
  Muscle weakness (not neuro) | 0 | 1
  Myalgia | 7 | 4
  Nausea | 10 | 51
  Neutropenia/granulocytopenia | 25 | 61
  PRBC transfusion | 0 | 3
  Pancreatitis | 0 | 1
  Personality/behavioral change | 1 | 0
  Petechiae/purpura | 0 | 1
  Platelet transfusion | 0 | 5
  Pruritus | 1 | 3
  Rash/desquamation | 4 | 10
  Renal failure | 0 | 1
  Reportable adverse event, NOS | 1 | 1
  Respiratory infect w/ neutrop | 0 | 2
  Rigors/chills | 2 | 1
  SGOT (AST) increase | 18 | 7
  SGPT (ALT) increase | 32 | 8
  Seizures | 0 | 2
  Sensory neuropathy | 0 | 2
  Stomatitis/pharyngitis | 0 | 1
  Surgery-wound infection | 3 | 0
  Syncope | 2 | 0
  Thrombocytopenia | 1 | 50
  Thrombosis/embolism | 1 | 1
  Typhlitis | 0 | 1
  Vertigo | 1 | 0
  Vomiting | 9 | 37
  Weakness (motor neuropathy) | 1 | 2
  Weight loss | 3 | 0

ADVERSE EVENTS:
Time Frame: While the patient is on treatment until resolution of acute toxicities with maximum grade reported
Description: Regular investigator assessments are reported after each cycle of protocol treatment
Arm/Group | Interferon | Biochemotherapy
Serious Adverse Events (participants affected / at risk) | 2/193 | 4/185
Other Adverse Events (participants affected / at risk) | 132/193 | 144/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon (N=193) | Biochemotherapy (N=185)
Platelet transfusion (Blood and lymphatic system disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Reportable adverse event, NOS (General disorders) | 1 | 0
Respiratory infect w/ neutrop (Infections and infestations) | 0 | 1
Cerebrovascular ischemia (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon (N=193) | Biochemotherapy (N=185)
Anemia (Blood and lymphatic system disorders) | 15 | 27
Diarrhea without colostomy (Gastrointestinal disorders) | 13 | 0
Nausea (Gastrointestinal disorders) | 37 | 67
Vomiting (Gastrointestinal disorders) | 23 | 52
Fatigue/malaise/lethargy (General disorders) | 79 | 27
Fever without neutropenia (General disorders) | 23 | 24
Rigors/chills (General disorders) | 27 | 0
Alkaline phosphatase increase (Investigations) | 0 | 16
Creatinine increase (Investigations) | 0 | 13
Leukopenia (Investigations) | 30 | 42
Neutropenia/granulocytopenia (Investigations) | 38 | 65
SGOT (AST) increase (Investigations) | 42 | 20
SGPT (ALT) increase (Investigations) | 53 | 20
Thrombocytopenia (Investigations) | 15 | 58
Weight loss (Investigations) | 12 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 11
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 35
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 23 | 14
Headache (Nervous system disorders) | 17 | 0
Anxiety/agitation (Psychiatric disorders) | 12 | 10
Depression (Psychiatric disorders) | 31 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 11
Hypotension (Vascular disorders) | 0 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No